CLINICAL TRIAL: NCT04088825
Title: Validation of the CONUT Software Tool for Screening Clinical Malnutrition in the University Hospital La Paz
Status: Completed | Type: Observational
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Other Study IDs: HULP PI-2340
Record Dates: First submitted 2019-09-12; First posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-08

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: CONUT screening system — CONUT has been working from june of 2010 and it has detected risk of malnutrition in 32% of the evaluated patients. The method collects information from databases of Admission Service (affiliation, age, date) and Laboratory (albumin, cholesterol, total lymphocytes) and generates, in the report of analytical results, "alert" information about each patient's nutritional risk and also nutritional recommendations based on the risk identified.

SUMMARY:
Nutrition Department of University Hospital La Paz decided to implement some method of screening in our centre which allowed us to detect as many patients with malnutrition risk as possible. Due to the large size of our centre, with about 1,500 beds and the few human resources in our unit, we chose to use the CONUT system (Nutritional Control), a 100% automatic method based on analytical parameters, very easy to use, low cost and whose validity is confirmed, characteristics that fulfilled our needs. The implementation of this nutritional screening method has led to a change in the ìnutritionafi culture of our centre respect to DRM in most of our professionals: doctors and nurses and even in the management team, so all of them understand the importance of the process and know about the available tools and knowledge to indicate an adequate and early nutritional support.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes
* Patients older than 15 years
* Patients admitted to the General Hospital or Traumatology area
* Patients who have signed the informed consent to participate in the study
* Patients who do not meet any exclusion criteria.

Exclusion Criteria:

* Pregnant women.
* Patients whose physical and / or psychic capacity prevents them from providing all the data collected by the evaluated methods or who do not have a caregiver.
* Non-collaborating patients in data collection
* Patients in whom a hospital stay of less than 48 hours is expected.
* Patients who at the time of performing the analyzes are in the ICU and OER

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Cross-sectional study in which the nutritional status of patients will be assessed in the first 72 hours of entry.
Sampling Method: Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2012-07-15 (Actual); Primary Completion 2012-09-15 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
To detect as many patients with malnutrition risk as possible | Three months
  The method collects information from databases of Admission Service (affiliation, age, date) and Laboratory (albumin, cholesterol, total lymphocytes) and generates, in the report of analytical results, "alert" information about each patient's nutritional risk and also nutritional recommendations based on the risk identified. Prior to its implantation several evaluations were performed in order to allow us to better know the extra workload, as it was the main factor that could limit our ability to assume that screening method and also many training activities for doctors and hospital health professionals who were increasingly assuming responsibilities in the nutritional treatment of their patients.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Gómez Candela, Msc, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Institute for Health Research IdiPAZ, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided